CLINICAL TRIAL: NCT07286435
Title: The Effect of Whole-Body Vibration Therapy Following Botulinum Toxin A Injection on Spasticity and Balance in Stroke Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Sevda Demir Türe, Specialist in Physical Medicine and Rehabilitation, Uludag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-16/7 and 09.09.2025
Record Dates: First submitted 2025-12-02; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Stroke Gait Rehabilitation
Keywords: stroke, whole body vibration, spasticity, balance; gait
MeSH Terms: conditions — Stroke; Muscle Spasticity

STUDY DESIGN:
Intervention Model Description: Single-center, randomized controlled, double-blind, prospective clinical trial
Who Masked: Participant, Investigator
Masking Description: The research assistant will conduct all outcome measurement assessments, and the researcher will be blinded to the type of program being administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The intervention group (Active Comparator): The intervention group will receive WBV program on a vibration platform in a semi-squat position for 10 minutes, 3 days a week for 4 weeks, with an amplitude of 4 mm and a frequency of 20Hz. This program will be administered using the 'Compex Winplate' device in the physical therapy room of our hospital's Department of Physical Medicine and Rehabilitation, under the supervision of a physical therapist. Both groups will be given a home exercise program consisting of calf muscle stretching and joint range-of-motion exercises, to be completed for 15 minutes per day, throughout the treatment period. The home program consists of stretching exercises for the ankle muscles, which can be performed without the use of additional materials. The participant will be given a pictorial guide after the physiotherapist explains the exercise program.
  Interventions: Device: Whole body vibration therapy
- The control group (Sham Comparator): The control group will receive sham WBV treatment (a vibration-free application) on a vibration platform in a semi-squat position for 10 minutes, three days a week, for four weeks. This program will be administered using the 'Compex Winplate' device in the physical therapy room of our hospital's Department of Physical Medicine and Rehabilitation, under the supervision of a physical therapist. Both groups will be given a home exercise program consisting of calf muscle stretching and joint range-of-motion exercises, to be completed for 15 minutes per day throughout the treatment period. The participant will be given a pictorial guide after the physiotherapist explains the exercise program.
  Interventions: Device: Sham whole body vibration therapy

INTERVENTIONS:
Device: Whole body vibration therapy — The intervention group will receive WBV program on a vibration platform in a semi-squat position for 10 minutes, 3 days a week for 4 weeks, with an amplitude of 4 mm and a frequency of 20 Hz. This program will be administered using the 'Compex Winplate' device in the physical therapy room of our hospital's Department of Physical Medicine and Rehabilitation, under the supervision of a physical therapist. Both groups will be given a home exercise program consisting of calf muscle stretching and joint range-of-motion exercises, to be completed for 15 minutes per day, throughout the treatment period. The home program consists of stretching exercises for the ankle muscles, which can be performed without the use of additional materials. The participant will be given a pictorial guide after the physiotherapist explains the exercise program.
  Arms: The intervention group
Device: Sham whole body vibration therapy — The control group will receive sham WBV treatment (a vibration-free application) on a vibration platform in a semi-squat position for 10 minutes, three days a week, for four weeks. This program will be administered using the 'Compex Winplate' device in the physical therapy room of our hospital's Department of Physical Medicine and Rehabilitation, under the supervision of a physical therapist. Both groups will be given a home exercise program consisting of calf muscle stretching and joint range-of-motion exercises, to be completed for 15 minutes per day throughout the treatment period. The participant will be given a pictorial guide after the physiotherapist explains the exercise program.
  Arms: The control group

SUMMARY:
The purpose of this clinical study is to evaluate the effect of Whole Body Vibration (WBV) therapy, applied two weeks after botulinum toxin type A (BoNT-A) injection, on spasticity and balance parameters in individuals with stroke who have ankle spasticity. The main questions it aims to answer are: Adjuvant WBV therapy administered after BoNT-A injection;

* Does it effectively improve spasticity?
* Is it an effective intervention for balance and walking functions? Researchers will compare the application of WBV to a placebo application (a vibration-free application) to evaluate the effect of adjuvant WBV therapy administered after BoNT-A injection on ankle spasticity, balance, and walking function in individuals with stroke.

DETAILED DESCRIPTION:
Materials and Methods:

Stroke participants who applied to the outpatient clinic of the Department of Physical Medicine and Rehabilitation at Uludağ University Faculty of Medicine and were evaluated at the rehabilitation council due to ankle spasticity, and for whom BoNT-A injection therapy was planned for the gastrosoleus muscles, will be evaluated for study eligibility. The study will include a total of 50 participants who meet the inclusion criteria. Participants to be included in the study will be randomly assigned to 2 groups, with 25 participants in each group, using computer-generated randomization. The study was planned as a prospective, double-masked, randomized controlled clinical study.

Informed consent will be obtained from participants who meet the inclusion criteria. Participants' demographic data (age, gender, height, and weight), stroke type (ischemic/hemorrhagic), side of hemiplegia (right/left), lesion location, comorbidities, pre-stroke functional status, and use of antispastic medication will be recorded.

For all participants who planned to receive BoNT-A injection therapy for ankle spasticity during outpatient clinic visits and who met the study criteria, 100-300 units of BoNT-A injection therapy will be administered to the gastrosoleus muscles by an experienced physical medicine and rehabilitation specialist. Thereafter, participants will be categorized into two groups of 25 individuals each based on a random number table.

* The intervention group will receive the WBV program on a vibration platform in a semi-squat position for 10 minutes, 3 days a week for 4 weeks, with an amplitude of 4 mm and a frequency of 20 Hz. This program will be administered using the 'Compex Winplate' device in the physical therapy room of our hospital's Department of Physical Medicine and Rehabilitation, under the supervision of a physical therapist.
* The control group will receive sham WBV treatment (a vibration-free application) for the same duration.

Both groups will be given a home exercise program consisting of calf muscle stretching and joint range-of-motion exercises, which will be completed for 15 minutes per day throughout the treatment period. The home program consists of stretching exercises for the ankle muscles, which can be performed without the use of additional materials. The participant will be given a pictorial guide after the physiotherapist explains the exercise program.

Study Algorithm: Power analysis was performed using the G*Power 3.1.9.6 program to calculate the sample size. The effect size of the difference between the two groups in terms of the Modified Ashworth Scale, VAS score, H-reflex, and Hmax/Mmax ratio was determined to be 0.80, with Chan et al.'s study serving as a reference. It was determined that at least 25 participants were required in each group to achieve 80% power and a significance level of 5%.

The data will be analyzed using IBM SPSS v. 25 statistical software. The obtained data will be analyzed and compared using appropriate statistical tests.

ELIGIBILITY:
Inclusion criteria:

* Participants with unilateral hemiparesis due to hemorrhage or infarction
* Participants aged 18-75 years
* Participants with MAS ≥2 spasticity in the ankle
* Participants with a Mini-Mental State Examination (MMSE) score of 24, indicating preserved cognitive and communication abilities
* Participants who can walk at least 100 meters with or without assistive devices
* Participants without joint contractures and with sufficient motor control to perform functional walking tests
* Participants who have not previously undergone vibration therapy

Exclusion Criteria:

* History of neurological disease (such as polyneuropathy or motor neuron diseases) other than a history of existing stroke
* History of recent fracture in the lower extremity
* Severe degenerative joint disease
* History of implants in the lower extremity or spine
* History of cardiac pacemakers
* Presence of uncontrolled hypertension and uncontrolled diabetes
* History of recent thromboembolism or infection
* Participants whose antispasmodic medication regimen was changed within 1 month prior to starting treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the maximum amplitude of the H-reflex, the Hmax/Mmax ratio, and F-wave parameters evaluated with EMNG. | "From enrollment to the end of treatment at 12 weeks"
  -ENMG evaluation: Initially (0), 2 weeks after BoNT-A injection (Week 2), at the end of WBV treatment (Week 6), and at Week 12, an experienced neurologist will perform EMG to assess ankle spasticity. The maximum amplitude of the H-reflex, the Hmax/Mmax ratio, and F-wave parameters will be measured and recorded
Change from Baseline in the static balance and postural stability assessment | From enrollment to the end of treatment at 12 weeks
  Initially (0), 2 weeks after BoNT-A injection (Week 2), at the end of WBV treatment (Week 6), and at Week 12, to assess static balance, participants will be evaluated for anteroposterior and mediolateral sway on both hard and foam surfaces with eyes open and closed using the HUR Smartbalance BTG4 balance platform (HUR-labs Oy, Kokkola, Finland). Additionally, limits of stability (LOS) measurements will be taken, and the results will be recorded.
MAS (Modified Ashworth Scale) | From enrollment to the end of treatment at 12 weeks
  MAS is a muscle tone assessment scale used to evaluate resistance during passive range of motion, requiring no instrumentation, and can be performed quickly. The scale is graded as follows: 0: No increase in muscle tone 1: Slight increase in muscle tone with catching and release or minimal resistance at the end of the range of motion when the affected part(s) are moved in flexion or extension 1+: Slight increase in muscle tone, manifesting as catching, followed by minimal resistance (less than half) for the remainder of the range of motion. 2: There is a marked increase in muscle tone throughout most of the range of motion, but the affected part(s) can still be moved easily. 3: Significant increase in muscle tone, difficulty with passive movement. 4: Affected part(s) fixed in flexion or extension
TUGT (Timed Up and Go Test) | From enrollment to the end of treatment at 8 weeks
  This Test assesses mobility; a chair and a stopwatch are required. The Test is conducted with the participant wearing their regular shoes, and they are allowed to use walking aids if necessary. A 3-meter area is designated in front of the chair. The participant is asked to stand up from the chair, walk a certain distance, and then sit down again. Time will tell the results of the Test.
Berg Balance Scale (BBS) | From enrollment to the end of treatment at 12 weeks
  It is used to assess functional balance and determine fall risk. The Test consists of 14 items. Values between 0 and 4 are given for each item. While 0 represents the worst value, 4 represents the best value. Four points indicate the ability to complete the task independently. The highest score is 56. Scores between 0-20 indicate balance impairment, scores between 21-40 indicate acceptable balance, and scores between 41-56 indicate good balance.

SECONDARY OUTCOMES:
The Functional Independence Measure (FIM) | From enrollment to the end of treatment at 12 weeks
  The Functional Independence Measure (FIM): indicates an individual's level of independence in daily life activities. It consists of 18 items, including sections on self-care, sphincter control, transfer, mobility, communication, social perception, and cognitive status, with a scoring range of 18-126. It consists of motor (13 items) and cognitive (5 items) subscales. All items will be answered using a 7-point Likert scale. A validity and reliability study in Turkish has been conducted.
The Visual Analog Scale (VAS) | From enrollment to the end of treatment at 12 weeks
  The Visual Analog Scale (VAS): is scored between 0 and 10. 0 represents the absence of spasticity during ambulation, and 10 represents the maximum intensity of spasticity that prevents ambulation.
10 m Walk Test | From enrollment to the end of treatment at 12 weeks
  10 m Walk Test: During the Test, the participant walks at a normal walking speed between two markers 10 meters apart, and the time taken is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Sevda Demir Ture, Principal Investigator — Uludag University; Alev Alp, Principal Investigator — Uludag University; Emel Oguz Akarsu, Principal Investigator — Uludag University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Picelli A, Santamato A, Chemello E, Cinone N, Cisari C, Gandolfi M, Ranieri M, Smania N, Baricich A. Adjuvant treatments associated with botulinum toxin injection for managing spasticity: An overview of the literature. Ann Phys Rehabil Med. 2019 Jul;62(4):291-296. doi: 10.1016/j.rehab.2018.08.004. Epub 2018 Sep 13. PMID 30219307
- [Background] Paoloni M, Giovannelli M, Mangone M, Leonardi L, Tavernese E, Di Pangrazio E, Bernetti A, Santilli V, Pozzilli C. Does giving segmental muscle vibration alter the response to botulinum toxin injections in the treatment of spasticity in people with multiple sclerosis? A single-blind randomized controlled trial. Clin Rehabil. 2013 Sep;27(9):803-12. doi: 10.1177/0269215513480956. Epub 2013 Mar 29. PMID 23543344
- [Background] Chan KS, Liu CW, Chen TW, Weng MC, Huang MH, Chen CH. Effects of a single session of whole body vibration on ankle plantarflexion spasticity and gait performance in patients with chronic stroke: a randomized controlled trial. Clin Rehabil. 2012 Dec;26(12):1087-95. doi: 10.1177/0269215512446314. Epub 2012 Oct 3. PMID 23035004